CLINICAL TRIAL: NCT01619670
Title: A Prospective Single Center Within Subject Controlled Observational Study to Evaluate Apligraf(R) in Nonhealing Wounds of Subjects With Epidermolysis Bullosa
Brief Title: A Observational Study to Evaluate Apligraf(R) in Nonhealing Wounds of Subjects With Epidermolysis Bullosa
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKBB 235/11
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Epidermolysis Bullosa; Wound Healing
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no intervention (No Intervention): standard wound care
- Apligraf (Active Comparator): non adhesive layer with apligraf
  Interventions: Device: Apligraf

INTERVENTIONS:
Device: Apligraf — non adhesive layer
  Arms: Apligraf

SUMMARY:
Epidermolysis Bullosa (EB) is a very rare disease, with a severe impact on the life of the patient and the caregiver. Epidermolysis Bullosa (EB) comprises a group of genetically determined skin fragility disorders characterized by blistering of the skin and mucosae following mild mechanical trauma. There is no specific proven treatment for any form of EB, and the mainstay of clinical management is based on protection and avoidance of provoking factors. Chronic nonhealing erosions and ulcers have been treated with conventional split-thickness skin grafts. Alternatively some patients may benefit from the use of autologous or allogeneic cultured keratinocyte grafts.

DETAILED DESCRIPTION:
Apligraf is a living bilayered cell therapy product. Apligraf is constructed of Type I bovine collagen. The mechanism of action of Apligraf is still unknown. No clinical evidence of rejection of Apligraf was observed when placed on acute or chronic wounds. Apligraf has been suggested to act as a "smart" material for wound healing by interacting with the surrounding environment to promote healing. It provides components with multiple actions, interacts with wounds in biological and physical ways, and appears to adapt to the wound environment and probably produces numerous pro-healing cytokines. The purpose of this study is to evaluate the use of Apligraf for the treatment of nonhealing wounds in subjects with epidermolysis bullosa. Apligraf will be evaluated for efficacy and safety compared to a conventional nonadherent dressing. The study is a pivotal, single center, within subject controlled observational trial in which the rate of wound healing, recurrence of EB lesions, subject report of pain will be compared to wounds treated with Control treatment. Subjects between 2 and 65 years of age, inclusive, with epidermolysis bullosa lesions will be screened for this study. For each subject at least two designated treatment sites will be selected. In case of two comparable treatment sites the most right side will receive Apligraf and the most left side will receive control. Efficacy will be assessed by clinical observations, wound tracings and photographs.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 2 and 65 years of age.
2. Subject with clinical confirmed diagnosis of EB.
3. Subject has at least two lesions, if in a situation with two non-adjacent EB lesions, at least 4 cm apart.
4. Subject with EB lesions at least 2 cm2 present for at least 3weeks. For the purposes of this study, a lesion is defined as a wound resulting from a post blister erosion.
5. Subject who is a female of child-bearing potential (females >10 years of age) must have a documented negative urine or serum pregnancy test. Sexually active females must be practicing a medically proven form of contraception during the course of the study period.
6. Subject or legal guardian must have read, understood and signed an institutional review board (IRB) approved Informed Consent Form or Assent Form.
7. Subject and/or legal guardian must be able and willing to follow study procedures and instructions.

   -

Exclusion Criteria:

* 1. Subject whose lesion has healed 20% or greater in area from post debridement (if applicable) Baseline Screen (Visit 1) to post debridement Day 0 (Visit 2) as determined by wound tracings.

  2. Subject with uncontrolled diabetes mellitus (glycosylated HbA1C > 10%), cancer (biopsy confirmed active malignancy), or positive HIV test.

  3. Subject is a child (<18 years of age) who is currently receiving or has received oral steroid therapy exceeding a total daily dose of 0.5mg/kg for more than two weeks, radiation or other immuno-suppressive therapy which would interfere with wound healing within the past four weeks.

  4. Subject is an adult (>18 years of age) who is currently receiving or has received chronic high dose steroid therapy exceeding a total daily dose of 20mg for more than two weeks, radiation or other immuno-suppressive therapy which would interfere with wound healing within the past four weeks.

  5. Subject who is currently on or has received topical steroidal therapy within 30 days before screening. Inhaled steroids are allowed.

  6. Subject with the presence of acute infections in the areas intended for treatment.

  7. Known hypersensitivity to bovine collagen or to the components of the Apligraf agarose shipping medium.

  8. Subject who is lactating or pregnant (hCG positive as determined by lab testing).

  9. Subject enrolled in any wound or investigational device study for any disease within the past four weeks.

  10. Subject who has received an investigational drug or biological treatment within three months.

  11. Subject with a history of alcohol or substance abuse within the previous year, which could interfere with study compliance such as inability to attend scheduled study visits or compliance with home dressing changes.

  12. Subject who, in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Proportion of wounds | through study week 12
  Proportion of wounds first achieving 100 % epithelialization of tissue with the absence of drainage (i.e. complete wound closure) through study week 12.

SECONDARY OUTCOMES:
Time | until 100% epithelialization
  Time until 100 % epithelialization of wound tissue with the absence of drainage (i.e.complete wound closure).

OTHER OUTCOMES:
Pain | Study duration
  Reduction of intensity of pain

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Arnold, MD, Principal Investigator — University Hospital Basel, Dep. Dermatology and Venereology, Basel/Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland